CLINICAL TRIAL: NCT05905354
Title: Clinical Study of HPV Therapeutic DNA Vaccine (NWRD08) in Patients With Cervical HPV16 and/or HPV18 Positive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newish Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NEWISH-HPV-001
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: HSIL of Cervix

STUDY DESIGN:
Intervention Model Description: 3+3 dose climb
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lose dose,high dose (Experimental): Four dose groups were set up: dose group 1, a single dose of 2mg, administered at week 0, 4 and 12, three times in total; Dose group 2, a single dose of 6mg, respectively at the 0, 4, 12 weeks, a total of 3 times; Dose group 3, a single dose of 2mg, was given at the 0, 2, 4, 12 weeks, a total of 4 times; Dose group 4, with a single dose of 6mg, was given 4 times at week 0, 2, 4 and 12, respectively. There were 3 subjects in each group. Climb from the low dose group to the high dose group.
  Interventions: Biological: NWRD08

INTERVENTIONS:
Biological: NWRD08 — Subjects in dose group 1 and 2 were intramuscularly injected with NWRD08 at week 0, week 4 and week 12 by electric pulse gene delivery instrument, respectively. Subjects in dose group 3 and 4 were intramuscularly injected NWRD08 at week 0, week 2, week 4 and week 12 by electric pulse gene delivery instrument, respectively.

SUMMARY:
This is an open-label exploratory clinical study. The main objective is to explore the immunogenicity of HPV therapeutic DNA vaccine NWRD08.

DETAILED DESCRIPTION:
The main objective is to explore the immunogenicity of HPV therapeutic DNA vaccine NWRD08.The secondary objective was to observe the safety of NWRD08 in cervical patients who were positive for HPV16 and/or HPV18, and to initially explore the efficacy of NWRD08.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. women who have sex;
3. HPV16 and/or 18 DNA and E6E7 mRNA were positive;
4. Patients with highly squamous intraepithelial lesions of the cervix confirmed by histology and cytology, or persistent cervical PV16 and/or 18 infection for more than 12 months;
5. Cervical tissue specimens/sections should be provided 4 weeks before the first treatment of HISL;
6. Electrocardiogram (ECG) is normal;
7. Women of reproductive age must have a negative serum pregnancy test within 1 week prior to the first dose and have agreed to use effective contraception during the study drug use period and within 6 months after the last dose of the study drug. For males, it should be surgical sterilization or consent to effective contraception during the study drug use period and within 6 months after the last study drug administration;
8. Have fully understood the study and voluntarily signed the ICF, be able to communicate well with the investigator and complete all treatments, examinations and visits required by the study protocol.

Exclusion Criteria:

1. any histopathologically confirmed adenocarcinoma in situ (AIS), high-grade vulvar, vaginal or anal intraepithelial tumors, or invasive cancers;
2. Patients with unsatisfactory colposcope;
3. Patients who were satisfied with colposcopy but not satisfied with ECC (patients who were positive for HPV18 or had abnormal adenocytes on cervical cytology but satisfied with colposcopy should undergo ECC examination);
4. Positive HPV type 31 or 33 or 45 or 52 or 58;
5. Have received cervical physical therapy;
6. pregnant, breastfeeding, or considering becoming pregnant during the study period;
7. previous history of therapeutic or preventive HPV vaccination;
8. Received any non-investigational inactivated vaccine injection within 2 weeks;
9. Received any non-investigational live vaccine within 4 weeks;
10. Acute or chronic bleeding or coagulopathy;
11. Less than two sites can be used for intramuscular injection;
12. Received chemotherapy, molecular targeted therapy, biological immunotherapy, or Chinese patent drugs for cervical lesions within 30 days before or during screening;
13. participated in other clinical trials within 30 days prior to screening, or was in the observation period of other clinical trials;
14. Continuous (more than 1 week) glucocorticoid therapy (dose equivalent to prednisone > 10 mg/ day), except hormone replacement therapy and endotracheal administration;
15. History of immune deficiency or autoimmune disease (such as rheumatoid joint disease, systemic lupus erythematosus, multiple sclerosis, etc.);
16. with uncontrolled severe infection;
17. Patients with a history of hepatitis B virus (HBV), hepatitis C virus (HCV) infection or human immunodeficiency virus (HIV) infection or syphilis carriers;
18. Patients with severe other organ dysfunction or cardiopulmonary disease, including myocardial infarction, stroke, congestive heart failure, severe lung disease, metabolic diseases, wound healing abnormalities, ulcers or fractures;
19. Epilepsy accompanied by medication (such as steroids or antiepileptic drugs);
20. Previous or present malignant neoplasms;
21. A history of severe allergies, or a history of allergic diseases, or an allergic constitution, or a severe iodine contrast allergy, meeting any of these criteria;
22. serious mental disorders;
23. A history of drug or alcohol abuse;
24. A pregnant or lactating woman, or a woman of childbearing age who has a positive blood pregnancy test, or a patient of childbearing age and her spouse who is unwilling to take effective contraceptive measures during the clinical study period and within 6 months after the end of treatment;
25. Patients deemed unsuitable for this clinical trial by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV 16/18 E6E7 specific immune response in peripheral blood after vaccination compared to before vaccination. | Week36
  Analysis of immunogenicity data included the level, type, subtype, and time and duration of specific humoral and cellular immune responses in peripheral blood before and after vaccination.

SECONDARY OUTCOMES:
Adverse Events (AEs) | End of study
  Adverse Events (AEs), adverse events according to type, frequency, severity [according to the Classification Scale of Adverse Events in Clinical Trials for Preventive Vaccines issued by the Center for Drug Evaluation (CDE) of the National Medical Products Administration in 2019], occurrence time, and severity. And whether it's related to treatment.
proportion of patients with HPV virus clearance | Week 36
  Proportion of patients with negative HPV16/18 DNA and E6E7 mRNA.
proportion of patients with regression of cervical lesions | Week 36
  1. HSIL patients 36 weeks group / 18 DNA and E6E7 mRNA overcast and histological ratio dropped below CIN1 and patients;
  2. HSIL patients 36 weeks group / 18 DNA and E6E7 mRNA overcast and histological the proportion of patients with squamous intraepithelial lesions;
  3. LSIL patients 18 DNA and 36 weeks group/E6E7 mRNA overcast and cytology squamous intraepithelial lesions;

CONTACTS AND LOCATIONS:
Overall Officials: Sun Guodong, Master, Principal Investigator — Shandong Heze Municipal Hospital
Locations (1):
- Heze Municipal Hospital, Heze, Shandong, China

IPD SHARING:
Plan to Share IPD: No